CLINICAL TRIAL: NCT04687371
Title: The Effect of Proprioseptive Vestibular Rehabilitation on the Balance, Functional Mobility, Posture, Sensory Profile and Quality of Life in Patients With Vertigo Due to Peripheral Vestibular Hypofunction
Brief Title: The Effect of Proprioseptive Vestibular Rehabilitation in Patients With Peripheral Vestibular Hypofunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Burcu Talu, Associate Professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020/190
Record Dates: First submitted 2020-12-18; First posted 2020-12-29 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2021-02

CONDITIONS: Vertigo, Peripheral; Vestibular Disease
Keywords: Vertigo; Peripheral Vestibular Hypofunction; Exercises; Balance; Functional Mobility; Quality of Life
MeSH Terms: conditions — Vertigo; Vestibular Diseases; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Experimental, Randomized Controlled Study
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Grup I (Experimental): Proprioceptive vestibular rehabilitation exercises, Cawthorne Cooksey Exercises and Gaze Stabilization exercises,
  Interventions: Other: Proprioceptive vestibular exercise
- Grup II (Experimental): Cawthorne Cooksey Exercises and Gaze Stabilization exercises
  Interventions: Other: Standard vestibular rehabilitation exercises
- Grup III (Other): No intervention will be made, patients will be asked to continue their daily life
  Interventions: Other: Controlled

INTERVENTIONS:
Other: Proprioceptive vestibular exercise — To assess effects of proprioceptive vestibular exercises training in patients with peripheral vestibular hypofunctions
  Other Names: Cawthorne cooksey exercises; Gaze stabilization exercises
  Arms: Grup I
Other: Standard vestibular rehabilitation exercises — To assess effects of standard vestibular rehabilitation exercises in patients with peripheral vestibular hypofunctions
  Other Names: Cawthorne Cooksey Exercises, Gaze Stabilization Exercises
  Arms: Grup II
Other: Controlled — First and last measurement will be taken. There will be no intervention. study will include 9 patients.
  Arms: Grup III

SUMMARY:
The aim of this study was to investigate the effect of proprioceptive vestibular rehabilitation on balance, functional mobility, posture, sensory profile and quality of life in patients with vertigo due to peripheral vestibular hypofunction.

DETAILED DESCRIPTION:
Peripheral vestibular system; It forms the part extending from the structures in the inner ear to the vestibular nuclei in the brainstem. Peripheral vestibular hypofunction is a chronic disease affecting one or both sides of the vestibular system, which occurs when the function of the vestibular organs, vestibular nerve, or both is reduced or destroyed. Many patients with peripheral vestibular hypofunction develop symptoms such as dizziness, vertigo, imbalance, gait disturbance. Many different exercise methods have been tried so far to relieve these symptoms and increase the functionality of the patient. In this study, we aimed to examine the effect of proprioceptive vestibular rehabilitation on balance, quality of life, posture, sensory profile and functional mobility in patients with vertigo due to peripheral vestibular hypofunction aged 18-65 years. Patients with vertigo due to peripheral vestibular hypofunction between the ages of 18-65 will be included in our study. The population of the research will be created by the cluster sampling method and the randomization of the patients to be recruited will be determined using the "research ramdomizer" computer program; Patients will be divided into 3 groups as experimental and control groups. A randomized controlled, single-blind study will be planned. Group I (experiment): Glance stabilization exercises, Cawthorne Cooksey Exercises and Proprioceptive vestibular rehabilitation exercises, Group II (experiment): Glance stabilization exercises and Cawthorne Cooksey Exercises and Group III (control): no exercise will be given, they will be asked to continue daily life. Exercises will be applied to each group for 8 weeks, 4 days a week, 30 minutes, in the presence of 1 set of physiotherapists and as a home exercise program every day of the week. Individuals will be evaluated before and 8 weeks after the treatment. Tinetti Balance Test for balance assessment, One leg stand test; timed up and go test for functional mobility assessment; Dizziness Disability Inventory for quality of life; mobile posture assessment application for posture assessment; Adult / Adolescent Sensory profile will be used for sensory assessment. Pre- and post-treatment and intergroup evaluations will be compared, and the effectiveness of proprioceptive vestibular rehabilitation on balance, functional mobility, posture, sensory profile and quality of life, and its superiority over standard exercises will be interpreted.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-65 years
* Diagnosis of vertigo according to the clinical examination performed by an Otorhinolaryngologist, Vestibular Evoked Myogenic Potentials (VEMP), Video Head Impulse Test (VHIT)
* Patients with Unilateral Peripheral Hypofunction
* After giving detailed information about the research, agreeing to participate in the study.

Exclusion Criteria:

* Severe hearing / vision impairment-loss
* Patients with neurological, orthopedic, circulatory system problems that may cause vertigo, dizziness and balance disorders
* Having severe hypertension / diabetes
* Previous participation in a vestibular rehabilitation program
* Being healthy
* Patients using drugs that may affect the treatment negatively
* Refusing to participate in a clinical trial
* Patients who cannot adapt to the training program
* Patients who discontinued their treatment
* Patients with different diagnoses that may disrupt the treatment during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Dizziness handicap inventory | 8 weeks
  It used to assess the quality of life in patients with vertigo
Tinetti balance test | 8 weeks
  It used to asses the balance (questionnaire, score)
Time up and go test | 8 weeks
  It used to assses the functionality (sec)
Adolescent/Adult Sensory Profile | 8 weeks
  In the test, 6 different sensory processing processes are evaluated. Includes assessments of taste/smell process, movement process, visual processing, touch process, activity level and auditory processing. Each item is scored with likert measurements between 1 and 5 points determined by the person.
Mobile application for Posture Analyze | 8 weeks
  It used to assess Posture (Degree)

CONTACTS AND LOCATIONS:
Overall Officials: Burcu TALU, Assoc. Prof., Principal Investigator — Inonu University
Locations (1):
- Inonu University, Malatya, Battalgazi/MALATYA, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozaltin GE, Talu B, Bayindir T. The effect of proprioceptive vestibular rehabilitation on sensory-motor symptoms and quality of life. Arq Neuropsiquiatr. 2024 Nov;82(11):1-10. doi: 10.1055/s-0044-1790568. Epub 2024 Sep 24. PMID 39317226